CLINICAL TRIAL: NCT02911805
Title: Bridging Animal and Human Models of Exercise-induced Visual Rehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: C1924-P
Record Dates: First submitted 2016-09-08; First posted 2016-09-22 (Estimated); Results first posted 2025-03-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Vision Disorders
Keywords: Exercise; Retinal Degeneration; Neuropharmacology; Brain-Derived Neurotrophic Factor; Biometry; Immunochemistry; Molecular Biology; Neurosciences; Ophthalmology
MeSH Terms: conditions — Vision Disorders; Motor Activity; Retinal Degeneration | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic Exercise (Active Comparator): Exercise 3 times a week
  Interventions: Behavioral: Aerobic exercise
- Balance Training (Placebo Comparator): Group balance training 3 times a week
  Interventions: Behavioral: Balance exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — Stationary bicycle ergometer @ 50-80% of maximal heart rate reserve for 20 minutes to 45 minutes
  Arms: Aerobic Exercise
Behavioral: Balance exercise — Instructor-led exercises done in a group setting for strengthening, balance, flexibility
  Arms: Balance Training

SUMMARY:
This study will determine whether blood biomarker changes predict sight-saving benefits of exercise.

DETAILED DESCRIPTION:
Investigators of the Atlanta VA Center for Visual and Neurocognitive Rehabilitation (CVNR) find a very high prevalence of blinding diseases in the aging Veteran population. There are few treatments for the disorders that threaten our Veterans' eyesight. The work proposed here is the first step in determining whether exercise can be used by aging Veterans as an inexpensive and self-controlled therapy for vision loss. In order to translate exercise therapy for vision into the clinic, the investigators need to identify biomarkers that can be used to predict visual benefits.

Though human and animal studies show that aerobic exercise is beneficial to specific central and peripheral nervous system functions, effects on the retina and vision were unknown until the investigators recently discovered that treadmill exercise directly protects retinal neurons in mice undergoing light-induced retinal degeneration (LIRD). The investigators found that exercise increased levels of brain-derived neurotrophic factor (BDNF) a blood protein in the blood, brain and eyes, whereas treatment of mice with a BDNF inhibitor prevented the protective effects of exercise.

For this study, the investigators will assess visual outcomes and serum biomarkers (e.g, BDNF) in 60 subjects age 18-89 before, during, and after aerobic exercise. Subjects currently enrolled in a 12-week study (under Institutional Review Board (IRB) 56726) examining the effects of aerobic exercise on cognition will have visual testing (ERG, visual acuity, contrast sensitivity, and OCT) and blood collection prior to, during and after the standardized 12-week aerobic exercise regimen to determine whether circulating biomarker levels and visual outcomes are correlated and whether biomarker levels are altered as predicted in animal studies.

This study will determine whether biomarker changes predict sight-saving benefits of exercise. As opposed to surgery or pharmacological treatments, exercise programs provide a means for Veterans to exert some control over their visual disease progression and will increase their overall health.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Aged 18 to 89
* Sedentary as defined by < 120 min/week of aerobic exercise over prior 3 months
* Non-demented (MMSE 24)

Exclusion Criteria:

* Severe diabetes requiring insulin
* Cognitive-executive function deficit (MoCA < 26)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2028-01-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Boatright, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aerobic Exercise | Balance Training
Started | 6 | 8
Completed | 6 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Balance Training | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 6 | 8 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (8.6) | 73.1 (4.0) | 73.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity - Mean Acuity Change
Description: Early Treatment Diabetic Retinopathy Study (ETDRS) chart was used. Higher scores mean a better outcome. The number of correct responses (e.g., number of letters read correctly) from a subject assessed prior to start of the first session of the the 12 week study was subtracted from the number of correct responses elicited at the end of the last session of the study. The means of these differences for each study group (Balance Training vs Aerobic Exercise) were compared by two-tailed t-test.
Time Frame: 12 weeks
Population: As per baseline analysis population description.
Measure: Mean (Standard Deviation); unit: Letters read correctly
Arm/Group | Aerobic Exercise | Balance Training
Number analyzed (Participants) | 6 | 8
Letters read correctly | 7.333 (8.501) | -4.875 (10.58)
Statistical Analysis 1: Comparison: Aerobic Exercise vs Balance Training; Test type: Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Contrast Sensitivity
Description: Contrast sensitivity: The contrast sensitivity of the subjects will be measured with the Pelli-Robson Chart or Contrast Sensitivity Chart following the instructions provided with the chart. The two sides of the Pelli-Robson Chart have different letter sequences but are otherwise identical. The chart should be illuminated as uniformly as possible, so that the luminance of the white areas is between 80 and 120 cd/ m2 with no glare. The patient should sit directly in front of the chart at a distance of 1 meter (use the same 1 meter string as for visual acuity testing to measure the eye-to-chart distance). Subjects should be prevented from seeing the chart until the contrast sensitivity testing actually begins. Subjects should wear their best distance correction.
Time Frame: 12 weeks
Reporting Status: Not Posted, anticipated posting 2027-12

3. Secondary Outcome: Concentration of Brain-Derived Neurotrophic Factor (BDNF) in Serum.
Description: Blood will be drawn prior to and after exercise sessions. From this, serum levels of brain derived neurotrophic factor (BDNF) will measured by immunoenzymatic assay.
Time Frame: 12 weeks
Reporting Status: Not Posted, anticipated posting 2027-12

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, did not differ from the definitions provided at this website.
Arm/Group | Aerobic Exercise | Balance Training
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT02911805/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT02911805/ICF_001.pdf